CLINICAL TRIAL: NCT07318480
Title: Cognitively-enhanced tDCS of the Dorsolateral Prefrontal Cortex to Reduce Craving in Cocaine Addiction
Brief Title: Transcranial Direct Current Stimulation (tDCS) for Treatment of Cocaine Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Soterix Medical (Industry)
Responsible Party: Principal Investigator, Rita Goldstein, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 23-1756; R01DA060914 (NIH)
Record Dates: First submitted 2026-01-01; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Cocaine Use Disorder; Cocaine Dependence; Substance Use Disorder (SUD)
Keywords: Transcranial Direct Current Stimulation (tDCS); Brain Stimulation; cocaine use disorder; drug craving; neuromodulation; neuroimaging
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Active tDCS with Cognitive Reappraisal (CR) (Experimental): Active Transcranial Direct Current Stimulation (tDCS) (Soterix Medical mini-CT tDCS stimulator), and Cognitive Reappraisal (CR)
  Interventions: Device: Transcranial Direct Current Stimulator (tDCS); Behavioral: Cognitive Reappraisal Training
- Active tDCS (Experimental): Active Transcranial Direct Current Stimulation (tDCS), (Soterix Medical mini-CT tDCS stimulator)
  Interventions: Device: Transcranial Direct Current Stimulator (tDCS)
- Sham tDCS (Sham Comparator): Sham (Placebo) Transcranial Direct Current Stimulation (tDCS), (Soterix Medical mini-CT tDCS stimulator)
  Interventions: Device: Transcranial Direct Current Stimulator (tDCS)
- Sham tDCS with Cognitive Reappraisal (CR) (Experimental): Sham (Placebo) Transcranial Direct Current Stimulation (tDCS) (Soterix Medical mini-CT tDCS stimulator), and Cognitive Reappraisal (CR)
  Interventions: Device: Transcranial Direct Current Stimulator (tDCS); Behavioral: Cognitive Reappraisal Training

INTERVENTIONS:
Device: Transcranial Direct Current Stimulator (tDCS) — Participants will have two electrodes applied (one anode, one cathode) administering active (real) or sham (placebo, not real) tDCS stimulation of the dorsolateral prefrontal cortex.
  Stimulation will last 20 minutes per day, three days per week, for 5 weeks
  Other Names: Soterix Medical mini-CT tDCS stimulator
Behavioral: Cognitive Reappraisal Training — Cognitive reappraisal of drug cues during stimulation sessions
  Arms: Active tDCS with Cognitive Reappraisal (CR); Sham tDCS with Cognitive Reappraisal (CR)

SUMMARY:
The researchers will test whether cognitively enhanced transcranial direct current stimulation (tDCS) of the dorsolateral prefrontal cortex can reduce craving in inpatients with cocaine use disorder. Neuroimaging before and after stimulation will establish the neural correlates of recovery and allow predictions of outcomes, which will be assessed throughout the study and one month after its completion. Results could pave the way towards development of a new self-administered intervention to reduce craving when it is needed the most, enhancing recovery real-time and in the natural environment in people with cocaine addiction as generalizable to other drugs of abuse and other disorders of self-control.

DETAILED DESCRIPTION:
Over the past decade, the US has been affected by a re-emerging stimulant use public health crisis and alarming increases in crack/cocaine-related overdose deaths. In contrast to other types of addiction, there are no FDA approved treatments for crack/cocaine use disorder (CUD). Developing and testing evidence-based treatment options for this population, and exploring the underlying neural substrates, are therefore urgently needed. Core symptoms of addiction are craving and heightened reactivity to drug cues, attributed to impairments in prefrontal functions. This study builds upon Phase-1 and Phase-2 trials testing whether transcranial direct current stimulation (tDCS) targeting the dorsolateral prefrontal cortex can reduce craving in treatment-seeking inpatients with CUD. Participants will be randomized to receive real or sham tDCS, combined with cognitive reappraisal training of drug cues or a control condition, in a double-blind, factorial design (N=120). Craving and drug use outcomes will be assessed throughout the intervention and at one-month follow-up. Neuroimaging will be used to examine neural correlates of treatment response. Results may inform development of scalable, self-administered interventions to reduce craving and relapse risk in cocaine addiction.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and give informed consent
* Men and women 18-60 years of age.
* For women of childbearing potential, current use of a medically acceptable form of birth control
* DSM-5 diagnosis of stimulant use disorder with crack/cocaine as the drug of choice

Exclusion Criteria:

* Lifetime diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar I disorder, or delusional disorder as confirmed by the MINI or autism spectrum disorder as confirmed by medical history at the screening visit
* Current clinically significant or unstable medical conditions, including metabolic, endocrinological, oncological or autoimmune diseases, infectious diseases common in people with substance use disorders including Hepatitis B and C or HIV/AIDS; use of medications deemed exclusionary by the study team; or any laboratory value outside the reference range that the senior investigator team considers to be of clinical relevance
* Head trauma with loss of consciousness (>30 min)
* History of neurological or developmental disease of central origin including stroke, brain tumor or seizures, encompassing those symptoms associated with periods of drug withdrawal or abstinence
* Metal implants or devices that may be impacted by the electrical stimulation and additional MR contraindications
* Women of childbearing potential must use a medically acceptable birth control method during the study and will be asked to take a pregnancy urine test before exposure to tDCS (or MRI)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
fMRI blood-oxygenation level dependent (BOLD) signal | At baseline and immediately after 5 weeks of tDCS.
  Neuroimaging - Measure of fMRI blood-oxygenation level dependent (BOLD) signal in the dorsolateral prefrontal cortex before and immediately after 5 weeks of tDCS.
Change in Self-Reported Craving Score | At baseline, immediately after 5 weeks of tDCS, and 1 month after interventions.
  Changes in measures of craving cocaine craving on a 0-9 point scale in response to interventions, with high scores indicating higher craving.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Goldstein, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. Any purpose. Proposals should be directed to NARC@mssm.edu. To gain access, data requestors will need to sign a data access agreement.